CLINICAL TRIAL: NCT07316673
Title: A Prospective Randomized Clinical Trial Comparing a Fast Fix Enhanced Arthroscopic System Versus Conventional Arthroscopic Suturing for Temporomandibular Disc Repositioning in Internal Derangement: Clinical, Functional, and Surgical Outcomes
Brief Title: A Prospective Randomized Clinical Trial Comparing a Fast-Fix-Enhanced Arthroscopic System Versus Conventional Arthroscopic Suturing for Temporomandibular Disc Repositioning in Internal Derangement: Functional, Clinical, and Surgical Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wajmah Sayed Karim Al Sayed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fast-Fix-Enhanced Arthroscopic
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Joint Internal Derangement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast-Fix-Enhanced Arthroscopic Disc Repositioning (Experimental)
  Interventions: Procedure: Fast-Fix-Enhanced Arthroscopic
- Conventional Arthroscopic Suturing Disc Repositioning (Active Comparator)
  Interventions: Procedure: (Conventional Arthroscopic Suturing Disc Repositioning)

INTERVENTIONS:
Procedure: Fast-Fix-Enhanced Arthroscopic — Device: The FasT-Fix system is a medical device designed for an "all-inside" arthroscopic meniscal repair.
  Arms: Fast-Fix-Enhanced Arthroscopic Disc Repositioning
Procedure: (Conventional Arthroscopic Suturing Disc Repositioning) — Arthroscopic TMJ discopexy using conventional suturing
  Minimally invasive surgical intervention
  Arms: Conventional Arthroscopic Suturing Disc Repositioning

SUMMARY:
This prospective randomized clinical trial evaluates the effectiveness of a Fast Fix-enhanced arthroscopic system compared with conventional arthroscopic suturing for temporomandibular joint disc repositioning in patients with TMJ internal derangement. Patients are randomly allocated into two groups and assessed for functional improvement (maximum mouth opening), pain reduction, joint symptoms, and surgical performance outcomes over a 6-month follow-up period. The study aims to determine whether the Fast Fix-enhanced technique provides superior clinical, functional, and surgical outcomes compared to conventional arthroscopic suturing

ELIGIBILITY:
Inclusion Criteria.

* Age ≥ 18 years.
* Both sexes.
* Patients with TMJ internal derangement (disc displacement without reduction).
* Patients indicated for arthroscopic disc repositioning following failure of conservative management.

Exclusion Criteria

* Previous TMJ surgery on the affected joint.
* Rheumatoid arthritis, systemic inflammatory joint disease, or other TMJ pathology (tumor, fracture, infection)
* Severe degenerative joint disease (osteoarthritis grade V) or ankylosis.
* Patients are unable to comply with follow-up assessments or MRI evaluation.
* Patients with TMDS are secondary to malocclusion.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Functional improvement assessed by Maximum Mouth Opening (MIO) | Baseline (preoperative) to 6 months postoperatively (with assessments at 3 months and 6 months; primary endpoint at 6 months
  MIO is measured as the maximal interincisal distance (in millimeters) using a ruler or digital caliper, with the primary endpoint being the change from baseline to 6 months postoperatively.

SECONDARY OUTCOMES:
Clinical outcomes , Pain reduction assessed using the Visual Analogue Scale (VAS) • Improvement of joint symptoms, including clicking and tenderness. | Baseline (preoperative), 3 months, and 6 months postoperatively
  Pain intensity assessed using the 10-cm Visual Analogue Scale (VAS), where 0 represents no pain and 10 represents unbearable pain.
Joint Symptoms (Clicking and Tenderness) | Baseline (preoperative), 3 months, and 6 months postoperatively
  Clinical evaluation of TMJ joint sounds (clicking) and joint tenderness through physical examination and patient report.
Surgical outcomes Total surgical time recorded | Intraoperative (day of procedure only)
  Total surgical time recorded intraoperatively from incision to completion of disc fixation, measured in minutes
surgical outcomes Technical Feasibility | Intraoperative (day of procedure only)
  Surgeon's intraoperative assessment of the feasibility of disc fixation using the assigned arthroscopic technique.